CLINICAL TRIAL: NCT03663530
Title: Impact of Circadian Misalignment on Energy Balance Regulation
Brief Title: Circadian Misalignment and Energy Balance
Acronym: CM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AAAR9547
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Food intake; Energy expenditure; Body composition; Meal timing
MeSH Terms: conditions — Obesity | interventions — Meals

STUDY DESIGN:
Intervention Model Description: This is a 2-period crossover study in which sleep is identical in duration and timing but meals/food intake is varied relative to the sleep episode.
Masking Description: Participants will be masked to the true outcomes of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circadian misalignment (Experimental): Meals in this condition will be delayed by 4 hours relative to the circadian alignment condition. Food intake during this period will be from 1 PM to 11 PM.
  Interventions: Behavioral: Meal times
- Circadian alignment (Active Comparator): Meals in this condition will be aligned to the sleep episode. Food intake during this period will be from 9 AM to 7 PM.
  Interventions: Behavioral: Meal times

INTERVENTIONS:
Behavioral: Meal times — Meal times vary based on the arm: aligned or misaligned

SUMMARY:
Preliminary findings from the investigators' lab suggest that circadian misalignment, occurring when meals and sleep are mistimed from one another, alters resting state neuronal processing in areas relevant to food reward and interoception; supporting a role of sleep and meal misalignment, on energy balance regulation. No study has been done to disentangle the effects of sleep and meal timing on body weight regulation, independent of sleep duration. This study will provide information to guide messaging related to timing of meals and sleep that can be translated to individuals whose sleep follows unconventional times, such as shift workers and those with jetlag and social jetlag.

DETAILED DESCRIPTION:
The proposed study will test whether the misalignment of eating occasions to the sleep period influences health markers. The goal of the proposed study is to determine whether eating out of synchrony with sleep influences risk of chronic diseases. The proposed study has both mechanistic and translational objectives. First, the investigators will test whether eating late in the day will influence energy balance (hormones, energy expenditure, nutritional intakes). Next, they will observe how misaligned meals, relative to aligned meals, influence behavior. Overweight men and women will be recruited to participate in a 2-phase, crossover study, with constant sleep periods. Phases will only differ in the alignment of meals to the sleep period: aligned = meals starting 1 h after awakening; misaligned = meals starting 5 h after awakening. Mechanistic aims will be addressed from measurements taken after 3 and 14 d of the intervention. The translational aim will be addressed after a 4 wk free-living period following the prescribed meal times for each phase. This proposed study, which will manipulate meal timing, without affecting total sleep time, is important because it will provide information on the mechanism by which circadian misalignment influences health. As such, the proposed study will be a stepping-stone in the establishment of lifestyle recommendations or therapies to personalize chronotype to reduce the risk of chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* All racial and ethnic groups
* Body mass index 20-34.9 kg/m2
* Average sleep duration ≥7 hour/night, assessed during 2-week screening period
* Eat within 1 hour of awakening at least 5 days/week
* Midpoint of sleep at 4 AM or earlier

Exclusion Criteria:

* <10 nights of sleep <7 hour during the 2-week screening period
* Daytime napping
* Current or past sleep disorder (Sleep Disorders Inventory); Insomnia Severity Index Score >10
* Current or past psychiatric disorder, including eating disorders and seasonal affective disorder
* Any psychological or psychiatric disorder deemed to interfere with study outcomes
* Smoking (currently smoking any cigarettes or using tobacco products, e-cigarettes and vapes, or ex-smokers <3 years)
* Night and rotating shift work
* Travel across time zones within 4 wk of the study
* History of drug or alcohol abuse or excessive alcohol consumption (>3 drinks/day for men or 2 for women)
* Recent weight change (>5% gain or loss of body weight over past 3 months) or active participation in diet or weight loss program in previous 3 months; any weight loss procedure
* Pregnancy or <1 year post-partum
* Diagnosed sleep apnea or high-risk score on Berlin questionnaire (2 or more categories with positive score)
* Depression (score >13 on Beck Depression Inventory II) or taking anti-depressive medications
* Restless leg syndrome and circadian rhythm disorders
* Dementia or cognitive impairments
* Taking psychoactive or hypnotic medications
* Taking chronic analgesic or anti-inflammatory medications
* Having had gastrointestinal surgery, including gastric bypass surgery
* Restrained eating or abnormal scores on the Three Factor Eating Questionnaire
* Contraindications for magnetic resonance imaging scanning
* Hematocrit <30%
* Taking beta blockers, as this can interfere with melatonin secretion

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | Change over 2-week period
  Metabolic chamber
Body composition | Change over 4-week period
  Quantitative magnetic resonance
Nutritional intakes | 4 weeks
  3-day food records

SECONDARY OUTCOMES:
Task-based functional neuroimaging | Change over 2-week period
  Brain responses to food stimuli
Resting state functional neuroimaging | Change over 2-week period
  Functional neuroimaging
Appetite | 4 weeks
  Visual analog scales
Hormones | Change over 2-week period
  Leptin, ghrelin, peptide tyrosine tyrosine, glucagon-like peptide 1

OTHER OUTCOMES:
Circadian rhythms | Change over 2-week period
  Melatonin and cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be available for sharing with other investigators. Data sharing requests should be made in writing and sent directly to the investigator(s) who generated the data. The purposes for using shared data should be stated in the request, and the data can only be used for research purposes. Data sharing agreements should be developed and accepted by both parties before data sharing takes place. Protecting the rights and privacy of human subjects and maintaining the study participants' confidentiality will be the first priority of our data sharing plan. We plan to follow the HIPAA privacy rule for de-identification of a dataset before transferring data.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after results of the main aims from the final dataset have been accepted for publication.
Access Criteria: Our methods of data sharing include: mailing CD-ROM containing data or e-mailing data files directly to the requestors. Normally, our data files are available in Excel or SAS format. Other data file formats can also be requested. The study's Statisticians will assist in preparing the required data files for data sharing. fMRI data will be uploaded to a data file sharing repository for anyone to use. These data will be de-identified prior to release.

REFERENCES:
- [Derived] Boege HL, Wilson KD, Kilkus JM, Qiu W, Cheng B, Wroblewski KE, Tucker B, Tasali E, St-Onge MP. Higher daytime intake of fruits and vegetables predicts less disrupted nighttime sleep in younger adults. Sleep Health. 2025 Oct;11(5):590-596. doi: 10.1016/j.sleh.2025.05.003. Epub 2025 Jun 11. PMID 40506285